CLINICAL TRIAL: NCT06226974
Title: Acute Effects of Static Stretching on the Shoulder Joint Position Sense of Overhead Athletes: a Randomized Crossover Trial
Brief Title: Acute Effects of Static Stretching on the Shoulder Joint Position Sense of Overhead Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ESS/FSA-374/23-3
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Static Stretching; Joint Position Sense; Proprioception; Shoulder; Overhead Athletes
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Condition (No Intervention): 5-minute rest.
- Static Stretching of 30 seconds Condition (Active Comparator): Static stretching of 30 seconds of muscles around the shoulder of the dominant upper limb:
  * Shoulder extension - shoulder extension with the hand resting on a door;
  * Doorway stretch - horizontal abduction with the shoulder in 90º of abduction, the elbow in 90º of flexion and the forearm leaning against a door;
  * Shoulder flexion - arms above the head against a wall;
  * Cross-body stretch - maximal horizontal adduction of the arm, with the opposite hand holding the stretch;
  * Overhead triceps - arm above the head and elbow flexed, with the other hand pulling the elbow;
  * Internal Rotation 90° stretch - with the shoulder at 90º of flexion and the elbow at 90º of flexion, the opposite hand and forearm forces the internal rotation.
  Interventions: Other: Static Stretching
- Static Stretching of 90 seconds Condition (Active Comparator): Static stretching of 90 seconds of muscles around the shoulder of the dominant upper limb:
  * Shoulder extension - shoulder extension with the hand resting on a door;
  * Doorway stretch - horizontal abduction with the shoulder in 90º of abduction, the elbow in 90º of flexion and the forearm leaning against a door;
  * Shoulder flexion - arms above the head against a wall;
  * Cross-body stretch - maximal horizontal adduction of the arm, with the opposite hand holding the stretch;
  * Overhead triceps - arm above the head and elbow flexed, with the other hand pulling the elbow;
  * Internal Rotation 90° stretch - with the shoulder at 90º of flexion and the elbow at 90º of flexion, the opposite hand and forearm forces the internal rotation.
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Static Stretching — * Shoulder extension - shoulder extension with the hand resting on a door;
  * Doorway stretch - horizontal abduction with the shoulder in 90º of abduction, the elbow in 90º of flexion and the forearm leaning against a door;
  * Shoulder flexion - arms above the head against a wall;
  * Cross-body stretch - maximal horizontal adduction of the arm, with the opposite hand holding the stretch;
  * Overhead triceps - arm above the head and elbow flexed, with the other hand pulling the elbow;
  * Internal Rotation 90° stretch - with the shoulder at 90º of flexion and the elbow at 90º of flexion, the opposite hand and forearm forces the internal rotation.
  Arms: Static Stretching of 30 seconds Condition; Static Stretching of 90 seconds Condition

SUMMARY:
The purpose of the study is to investigate the acute effects of static stretching on the shoulder joint position sense of overhead athletes.

DETAILED DESCRIPTION:
A crossover randomized controlled trial will be conducted with 17 overhead athletes (9 males and 8 females). All of them will perform the 3 study conditions in random order: a control (5-minute rest), and static stretching of 30 or 90 seconds of muscles around the shoulder. The shoulder joint position sense will be assessed before and immediately after these conditions, and tested by active repositioning for the range of 110º of flexion, with a video camera. Absolute, relative and variable angular errors will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 30 years
* Competitive overhead athletes (basketball, handball, volleyball, swimming)
* Normal range of motion of flexion of the shoulder

Exclusion Criteria:

* History of injury of the shoulder joint in the previous 6 months
* Positive shoulder joint integrity tests (anterior drawer; fulcrum test; Jerk test; and sulcus sign)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Absolute angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The absolute value of the difference between the target range and the achieved range
Relative angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The arithmetic difference between the target range and the range achieved
Variable angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The standard deviation of the 3 repositionings

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior Saúde Fernando Pessoa, Porto, Portugal